

# Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy

**Study Protocol** 

(Pages 2 - 6)

#### **Study Protocol**

Study titled "Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy" was approved by Marmara University Faculty of Medicine Clinical Researches Ethics Committee meeting on 07.04.2017 with approval number: 09.2017.297 (Annex-1).

The legal representatives of the children who participated in the study were informed about the aim, duration and the programs to be applied throughout the study. Volunteer Information Form has been signed and approved in accordance with the standards deemed appropriate by the Clinical Researches Ethics Committee of Marmara University Faculty of Medicine (This form can be seen on Informed Consent Form (ICF) section). The study was conducted in accordance with the Declaration of Helsinki.

#### Hypothesis of the Study

H<sub>0</sub>: Addition of the exercises performed with Simulated Hypotherapy device to the neurodevelopmental (NDT) based rehabilitation program in children with cerebral palsy does not contribute positively in improving the efficiency of lower extremity functions, body control and spasticity.

H<sub>1</sub>: Addition of the exercises performed with Simulated Hypotherapy device to the neurodevelopmental (NDT) based rehabilitation program in children with cerebral palsy contributes positively to improve the efficiency of lower extremity functions, body control and spasticity.

#### Randomization of the Study Groups

Children with Cerebral Palsy who applied to the Bulgurlu Unimpeded Life Center for rehabilitation were invited to participate in the study. Children who volunteered to participate and whom met the criteria for participation were randomized with simple random sampling method and divided into two groups. Individual Neurodevelopmental (NDT) based rehabilitation programs were applied to the participants in Group I for 8 weeks. After 8 weeks of only Neurodevelopmental therapy (NDT) based rehabilitation, Simulated Hypotherapy system was added to the rehabilitation program, and the name of the was changed into Group II (the study group).

#### **Inclusion Criteria**

- Having a diagnosis of Spastic Cerebral Palsy,
- Children aged between 5 18 years,
- GMFCS level is I, II or III,
- Independent seating
- Walking at least 10 meters independently,
- Can understand simple verbal instructions,
- Those with a spasticity level less than 2 according to MAS,
- Having bilateral hip abduction enough to sit on the hippotherapy device,
- Voluntary acceptance to participate in the study

#### **Exclusion Criteria**

- Having hip dislocation,
- Severe contracture or deformity,
- Scoliosis (above 20 degrees),
- Acute uncontrolled acute seizures,
- Epilepsy,
- Visual and auditory problems,
- Injection of botulinum toxin in the last 6 months,
- History of surgical operation such as muscle relaxation, tendon extension and selective dorsal rhizotomy in the last 6 months.

#### **Applied Evaluations**

Evaluations are applied three times: before treatment, in week 8 (end of NDT) and in week 16 (end of simulated hippotherapy training). All evaluation data are noted to 'Participants Tracking Form' (Annex-2). Primary outcome measures and applied evaluations are shown in Table 1.

**Table 1.** Primary outcome measures and applied evaluations

| Primary Outcome Measures | Applied Evaluations |
|---|---|
| Functional Level | Gross Motor Functional Classification<br>System (GMFCS) |

| Spasticity | Modified Ashworth Scale (MAS) |
|---|---|
| Range of Motion (ROM) | Goniometer |
| Gross Motor Function | Gross Motor Function Measure - 88 |
| Trunk Movements | Trunk Impairment Scale (TIS) |
| Functional Independence | The Functional Independence Measure for Children (WeeFim) |
| Balance | Pediatrics Balance Scale (PDS) |
| Soft Tissue Assessment | Myoton PRO® Device |
| Gait Analysis | FreeMed® |
| Balance in Daily Living Activities | Pedalo® Balance Device |

Functional level will be defined with 'Gross Motor Functional Classification System (GMFCS), spasticity with 'Modified Ashworth Scale', lower extremity joint range of motion (ROM) with 'goniometer', gross motor functions with 'Gross Motor Function Measure (GMFM-88)', the functional strength of the body, its postural control and the nature of the trunk movements with 'Trunk Impairment Scale', functional independency for activities in children with 'The Functional Indepence Measure for Children (WeeFim)', the balance with an assessment tool adapted from the Berg Balance Scale (BDS) for the children in daily living activities 'Pediatric Balance Scale (PDS)', superficial skeletal muscles, connective tissues such as tendons and ligaments and other soft tissues with 'Myoton®PRO Digital Palpation Device', gait analysis with 'FreeMed® (Sensör Medica)' and the balance during sitting and standing positions with 'Pedalo Balance Device'.

#### **Treatment Program**

The participants in the study will be rehabilitated in Bulgurlu Unimpeded Life Center twice a week for 16 weeks in total (Duration of one session is 45 minutes).

Group I (Control Group) will receive individual Neurodevelopmental (NDT) based rehabilitation program.

Group II (Study Group) will receive individual NDT based rehabilitation program (25 minutes) + Simulated Hippotherapy System (20 minutes).

#### **Simulated Hippotherapy System Training Protocol**

In addition to the 25-minute neurodevelopmental treatment program, a 20-minute simulated hippotherapy system will be used. Programs that can be controlled by software and prepared according to the needs of the participants will be used. The simulated horse will be directed to reveal the contraction in the desired area. It is aimed to increase the strength of the desired muscles and to improve the body control, relaxation of muscles. EMG will be used to monitor how the muscles respond to action.

#### Neurodevelopmental Therapy (NDT) Based Rehabilitation

In accordance with the needs of the patients for their gross motor functions, the children in both groups were included in the NDT program, which was determined according to the age, sex, mental status and preferences of the individual. NDT program will include; rehabilitation of muscle tonus disorders, sensory-perception-motor integrity enhancement, exercises to increase extremity functions and body control, stretching and strengthening exercises due to muscular tightness and weakness, exercises to accommodate movements in daily life, and training of activities such as standing up, walking, body care.

# Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy

**Statistical Analysis Plan (SAP)** 

(Pages 7 – 8)

#### **Statistical Analysis Plan (SAP)**

The statistical program Statistical Package for Social Sciences (SPSS) Version 11.5 (SPSS Inc., Chicago, IL, USA) will be used in the data analysis of the study. The p value of p<0.05 will be considered to be statistically significant in the data analysis. One sample Kolmogorov-Smirnov test will be used to investigate the appropriateness of the variables to normal distribution.

Intra-group analysis of the evaluation parameters that conform to the normal distribution will be done by Paired t-test and the intergroup analysis will be done by Independent t-test. Wilcoxon t-test will be used for intragroup analysis of parameters that do not comply with normal distribution, and Mann Whitney-U Test will be used for intergroup analysis.

# Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy

**Informed Consent Form (ICF)** 

(Pages 9 - 14)

February 28, 2019

#### **Informed Consent Form (ICF)**

#### **Description of the Physiotherapist**

This study, if you accept your child to be participated, is a scientific research and it is titled as "Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy". In this study, functional level will be defined with 'Gross Motor Functional Classification System (GMFCS), spasticity with 'Modified Ashworth Scale', lower extremity joint range of motion (ROM) with 'goniometer', gross motor functions with 'Gross Motor Function Measure (GMFM-88)', the functional strength of the body, its postural control and the nature of the trunk movements with 'Trunk Impairment Scale', functional independency for activities in children with 'The Functional Indepence Measure for Children (WeeFim)', the balance with an assessment tool adapted from the Berg Balance Scale (BDS) for the children in daily living activities 'Pediatric Balance Scale (PDS)', superficial skeletal muscles, connective tissues such as tendons and ligaments and other soft tissues with 'Myoton®PRO Digital Palpation Device', gait analysis with 'FreeMed® (Sensör Medica)' and the balance during sitting and standing positions with 'Pedalo Balance Device'. The study, which is planned to last in 16 weeks, requires participants to attend the study regularly for twice a week and each day for one session which is 45 minutes. There will be no disruption of the body during the process.

This research will be carried out by Neslihan KARABACAK, PT (Tel: +90 534 ), Canan Günay YAZICI, PT, MSc (Tel: +90 538 ) and will be under the supervision of Zübeyir SARI, PT, MSc, PhD, Assoc. Prof. at Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation.

Your child is being invited to a research project. It is very important for you to understand why and how this research will be done before making a decision. Please take some time and read the following informations carefully, discuss it with others if you wish. If you have an unclear section or need more detailed information, you can get information from us. You are invited to our research because we think your child matches the criterias to be included. We would like to note that participation is voluntary and that refusal to participate does not lead to any penalty or loss of any benefit. In the same way, you can withdraw from the research at any time.

After getting the demographic information of the participants, the upper extremity functions will be measured by the above physiotherapist and with the mentioned tests. The evaluation tests will be repeated 3 times throughout the treatment. The data obtained from the assessments will be recorded in the computer and the changes during pre- and post-treatment will be analyzed. The assessments applied to the participants in our research do not have any known harm. In the event of any unexpected damage in the evaluation process or during the rehabilitation process, the information will be given immediately to you. In case of any damage to the participants, the necessary applications shall be covered by the researchers without any recourse. For this, you will not be charged any fees, neither you nor your social security insurance.

While participation in the research does not help you immediately, it is hoped that our research results will have benefits for the organization, society or science in the future. You will not be charged any fees for the purposes of the research or for the social security institution to which you are affiliated.

#### **Consent of the Participant**

I have read the entire information form clearly and understood or because I do not know how to read/not able to or do not understand the language it was read or translated to me. I was given the opportunity to ask, evaluate and decide on my health status both during and after my application and when filling this form in. All kinds of treatment and diagnostic alternatives, including the possibility of not getting the treatment, their risks and dangers are explained.

| Name and the Surname of the Participant and Legal Representative: | |
|---|---|
| Data | Signatura |
| Date: | Signature: |
| Name and Surname of the Withness: | |
| Date: | Signature: |

#### **Declaration of the Physiotherapist**

I gave the patient the necessary information about the study and the procedures to be performed. I believe that the patient understood this information, asked me the questions that she/he wanted to ask, and accepted the process with her/his free will.

Researcher: Physiotherapist Neslihan KARABACAK

**Address:** Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation- Başıbüyük . Maltepe /Istanbul/TURKEY

Mobile Phone: +90 534 E-mail: neslikarabacak@gmail.com

Date: Signature:

Researcher: Physiotherapist Canan GÜNAY YAZICI

**Address:** Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation - Başıbüyük . Maltepe/Istanbul/TURKEY

Mobile Phone: +90 538 E-mail: cnngnyzc@gmail.com @gmail.com

Date: Signature:

#### **Declaration of the Participant / Legal Representative**

I understand that a medical research will be carried out and the above information about this research was explained to me. I know my child is invited to this research as a participant. If I participate in this research, I believe that the confidentiality of the information of my child during research will be treated with great care and respect. I was given enough information that my child's personal information would be protected with care during the use of the research and the results will only used for educational and scientific purposes. During the research I can withdraw my child from the study at any time without any cause (But in that case I am aware of the difficult situation it would cause to the reaseachers if I do not give any notice). I don't take any financial responsibility for the research expenses. There will be no payment for me. Whether directly, indirectly arised any health problem that may occur during the research, I will not undergo any monetary burden. When we encounter any health problem during the research; at any hour, I know I can call my physiotherapist. My child does not have to be participated in this research or may not participate. We have not experienced any compelling behavior to participate in the research. If we refuse to participate, I know that this will not bring any harm to our medical care and our relationship with my physiotherapist. I have understood all the explanations made to me in detail. At the end of a certain period of thinking on my own, I decided that my child could take part in this research project as a participant. On behalf of my child, I accept this invitation voluntarily.

I have read the text above which shows the information that should be given to the volunteer before investigating. These were written and was explained verbally. With these conditions, I agree to participate in this research without any pressure or compulsion on me and my child. A signed 2 copies of this form, which consists of 4 pages, a copy of the documents will be given to me.

| Name and the Surname of the Participa | ant and Legal Representative: |
|---|---|
| Date: | Signature: |
| Name and Surname of the Withness (whe end): | who have witnessed the process of receipt until |
| Date: | Signature: |

The researcher who made the explanations,

Researcher: Physiotherapist Neslihan Karabacak

Address: Marmara University, Institute of Health Sciences, Department of

Physiotherapy and Rehabilitation - Başıbüyük . Maltepe/Istanbul/TURKEY

**Mobile Phone:** +90 534 **E-mail:** neslikarabacak@gmail.com

Date: Signature:

Researcher: Physiotherapist Canan GÜNAY YAZICI

Address: Marmara University, Institute of Health Sciences, Department of

Physiotherapy and Rehabilitation - Başıbüyük . Maltepe/Istanbul/TURKEY

Mobile Phone: +90 538 E-mail: cnngnyzc@gmail.com @gmail.com

Date: Signature:

## Development of Simulated Hippotherapy System and Investigation of the Effectiveness in Children with Cerebral Palsy

Annex

(Pages 15 – 25)

February 28, 2019

# **Annex 1.** Marmara University Faculty of Medicine Clinical Researches Ethics Committee Approval (Approval made at the meeting on 07.04.2018 with number: 09.2017.297)



#### Marmara Üniversitesi Tıp Fakültesi Klinik Araştırmalar Etik Kurulu

| BAŞVURU<br>BİLGİLERİ | PROTOKOL KODU | 09.2017.297 |
|---|---|---|
| | PROJE ADI | Simüle Hippoterapi Sisteminin Geliştirilmesi ve Serebral<br>Palsi'li Çocuklarda Etkinliğinin Araştırılması |
| DILOILE KI | SORUMLU ARAŞTIRICI ÜNVANI/ADI | Doç. Dr. Zübeyir SARI |

| | Tarih 07.04.2017 | | | | | |
|---|---|---|---|---|---|---|
| | alınarak incelenmis ve gerçekl | ilen araştırma başvuru dosyası vi<br>leştirilmesinde sakınca bulunmad<br>k proje değişiklikleri (katılımcılar<br>tedir. | ığı için Kurulumı | ezen onaylane | masina oy bi | rliği ile karar verilmiştir. C |
| YELER | | | | | | |
| Unvam / Adı / Soyadı | Uzmanlık Dah | Kurumu / EK Üyeliği | Onaylanan Pro<br>ite İlişkisi | | dantiya<br>atilum | Imza |
| Prof.Dr. Haner DİRESKENEL | i Romatoloji | M.Ü Tıp Fakültesi/ Başkan | Var Yok | Evet | Hayır | 10 |
| Prof.Dr. Tillin ERGUN | Dermatoloji | M.Ü Tıp Fakültesi/Başkan<br>Yed. | Var Yok | Evet | Hayır | 8 |
| Prof. Dr. Sefik GÖRKEY | Tip Tarihi ve Etik | M.Ü Tıp Fakültesi/Üye | Var Yok | | Hayır | 2 Jan |
| Prof.Dr. Handan KAYA | Puteloji | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet | Hayır | 1 |
| Prof.Dr. M.Bahadır GÜLLÜO | GLU Genel Cerrahi | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet | Hayır | |
| Prof.Dr. Atila KARAALP | Farmakoloji | M.Ĉ Tip Fakiiltesi/Ĉye | Var Yok | Ever | Hayir | |
| Prof.Dr. Semra SARDAS | Eczaci | M.C Eczacilsk Fuk/Üye | Var Yok | Evet | Hayır | |
| Prof.Dr. Başak DOĞAN | Diş Hekimi | M.Ü Diş Hekimliği Fak⊅Üye | Var Yok | Evet | Hayır | |
| Prof. Dr. Beste Melek ATASOY | Radyasyon<br>Onkolojisi | M.C Tıp Fakültesi/Cye | Var Yok | Evet | Hayır | Ili |
| Dog. Dr. Elif KARAKOÇ AYD | INER Cocuk Sağlığı ve<br>Hastalıkları | M.C Tip Fakültesi/Cye | Var Yok | Evet | Hayır | Avo |
| Dog.Dr. Meltem KORAY | Diş Hekimi | İstanbul Üniv. Diş Hekimliği<br>Fak,/Üye | Var Yok | Evet | Hayır | |
| Doç. Dr. Gürkan SERT | Hukukçu | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet | Hayır | *() |
| Yrd.Doç.Dr: Figen DEMİR | Halk Sagligi | Acıbudem Üniv. Tıp Fak. | Var Yok | Evet | Hayır | |
| Yrd.Doç.Dr. Pınar Mega TİBEI | R Biyofizik | M.Ĉ Tip Fakültesi/Ĉye | Var Yok | Evet | Hayır | M |
| Gözde Aynur MİRZA | Sağlık Mensubu<br>olmayan kişi | Serbest | Var Yok | Evet | Hayır | yes - |

# **Annex 2. Participants Tracking Form**

| No. | | Date. | | |
|---|---|---|---|---|
| Name-Surname | | | | |
| Adress | | | | |
| Phone | | | | I |
| Gender | Female | Male | Age | |
| Height | | | Weight | |
| CP Type | Hemiparetic [ | Diparetic | Quadrij | paretic |
| GMFCS Level | I | II | l III | |
| Education Level | | | | |
| Having surgery/date | | | | |
| Botulinum toxin injections and date of apply | | | | |
| Auxiliary tool use | | | | |
| Orthesis / device use | | | | |
| History of any disease / trauma | | | | |
| Any drug use at the moment? | | | | |

# RANGE OF MOTION

| MEASURE | BEFORE | | WEEK 8 | | WEEK 16 | |
|-----------------------|--------|-------|--------|-------|---------|-------|
| | LEFT | RIGHT | LEFT | RIGHT | LEFT | RIGHT |
| Hip flexion | | | | | | |
| Hip extansion | | | | | | |
| Hip internal rotation | | | | | | |
| Hip external rotation | | | | | | |
| Hip abduction | | | | | | |
| Hip adduction | | | | | | |
| Knee flexion | | | | | | |
| Knee extansion | | | | | | |
| Dorsi flexion | | | | | | |
| Plantar flexion | | | | | | |

### **Modified Ashworth Scale**

| MEASURE | BEFORE | | WEEK 8 | | WEEK 16 | |
|---------------|--------|-------|--------|-------|---------|-------|
| | LEFT | RIGHT | LEFT | RIGHT | LEFT | RIGHT |
| Hip adduction | | | | | | |
| Hamstring | | | | | | |
| Gastrocnemius | | | | | | |
| Soleus | | | | | | |

## **Myoton®PRO Digital Palpation Device**

| MEASURE | BEFORE | | WEEK 8 | | WEEK 16 | |
|---------------|--------|-------|--------|-------|---------|-------|
| | LEFT | RIGHT | LEFT | RIGHT | LEFT | RIGHT |
| Hip flexion | | | | | | |
| Hip adduction | | | | | | |
| Hamstring | | | | | | |
| Quadriceps | | | | | | |
| Gastroknemius | | | | | | |
| Soleus | | | | | | |

## **Modified Ashworth Scale (Please mark)**

| Grade | Description |
|---|---|
| 0 | No increase in muscle tone |
| 1 | Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part/s is/are moved in flexion or extension. |
| 1+ | Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM. |
| 2 | More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. |
| 3 | Considerable increase in muscle tone, passive movement difficult. |
| 4 | Affected part(s) rigid in flexion or extension. |

ROM, range of motion.

## **Gross Motor Functional Classification System (GMFCS) (Please mark)**



# Trunk Impairment Scale (Please mark)

| Item | | | |
|---|---|---|---|
| 1 | Static sitting balance<br>Starting position | Patient falls or cannot maintain starting position for 10 seconds without arm support Patient can maintain starting position for 10 seconds If score = 0, then TIS total score = 0 | □ 0<br>□ 2 |
| 2 | Starting position Therapist crosses the unaffected leg over the hemiplegic leg | Patient falls or cannot maintain sitting position for 10 seconds without arm support Patient can maintain sitting position for 10 seconds | □ 0<br>□ 2 |
| 3 | Starting position Patient crosses the unaffected leg over the hemiplegic leg | Patient falls Patient cannot cross the legs without arm support on bed or table Patient crosses the legs but displaces the trunk more than 10 cm backwards or assists crossing with the hand Patient crosses the legs without trunk displacement or assistance | |
| | | Total static sitting balance | 17 |
| 1 | Dynamic sitting balance Starting position Patient is instructed to touch the bed or table with the hemiplegic elbow (by shortening the hemiplegic side and lengthening the unaffected side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 2 and 3 score 0 | □ 0<br>□ 1 |
| 2 | Repeat item 1 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 3 scores 0 | □ 0<br>□ 1 |
| 3 | Repeat item 1 | Patient compensates Possible compensations are: (1) use of upper extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur), (4) knee flexion, (5) sliding of the feet Patient moves without compensation | □ 0<br>□ 1 |
| 4 | Starting position Patient is instructed to touch the bed or table with the unaffected elbow (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 5 and 6 score 0 | □ 0<br>□ 1 |
| 5 | Repeat item 4 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 6 scores 0 | □ 0<br>□ 1 |

| 6 | Re | peat item 4 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femury (4) knee flexion, (5) sliding of the feet Patient moves without compensation | |
|---|---|---|---|---|
| 7 | Pai<br>hei | arting position<br>tient is instructed to lift pelvis from bed or table at the<br>miplegic side (by shortening the hemiplegic side and lengthenin<br>e unaffected side) and return to the starting position | Patient demonstrates no or opposite shortening/lengthening 1g Patient demonstrates appropriate shortening/lengthening 1f score = 0, then item 8 scores 0 | □ (<br>□ 1 |
| 8 | Re | peat item 7 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation | |
| 9 | Pai<br>un | arting position<br>tient is instructed to lift pelvis from bed or table at the<br>affected side (by shortening the unaffected side and lengthenir<br>e hemiplegic side) and return to the starting position | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 10 scores 0 | □ (<br>□ 1 |
| 1 | 0 Re | peat item 9 | Patient compensates. Possible compensations are: (1) use of upper extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation Total dynamic sitting balance | □ (<br>□ 1<br>/1( |
| 1 | Starti<br>Patier<br>shoul | dination ng position nt is instructed to rotate upper trunk 6 times (every shoulder d be moved forward 3 times), first side that moves must be elegic side, head should be fixated in starting position | Rotation is asymmetrical | □ 0<br>□ 1<br>□ 2 |
| 2 | Repea | at item 1 within 6 seconds | • | □ 0<br>□ 1 |
| 3 | Patier<br>shoul | ng position<br>at is instructed to rotate lower trunk 6 times (every knee<br>d be moved forward 3 times), first side that moves must be<br>elegic side, upper trunk should be fixated in starting position | Rotation is asymmetrical | □ 0<br>□ 1<br>□ 2 |
| 4 | Repea | at item 3 within 6 seconds | • | □ 0<br>□ 1<br>/6 |
| | | | Total Trunk Impairment Scale | /23 |

## **Pediatric Balance Test (Please mark)**

All items are scored between 0 and 4 and the total score is calculated.

| | Pediatric Balance Scale Items |
|-----------------------------------|----------------------------------------|
| 1 | Sitting to standing |
| 2 | Standing to sitting |
| 3 | Transfers |
| 4 | Standing unsupported |
| 5 | Sitting unsupported |
| 6 | Standing with eyes closed |
| 7 | Standing with feet together |
| 8 Standing with one foot in front | |
| 9 | Standing on one foot |
| 10 | Turning 360 degrees |
| 11 | Turning to look behind |
| 12 | Retrieving object from floor |
| 13 | Placing alternate foot on stool |
| 14 | Reaching forward with outstretched arm |

## The Functional Indepence Measure for Children (WeeFim) (Please mark)

| Items | Descriptive Items |
|----------------------|--------------------|
| Domain 1: self-care | |
| (maximum = 56) | |
| 1 | Eating |
| 2 3 | Grooming |
| 3 | Bathing |
| 4<br>5 | Dressing-upper |
| 5 | Dressing-lower |
| 6 | Toileting |
| 7 | Bladder |
| 8 | Bowel |
| Domain 2: mobility | |
| (maximum = 35) | |
| 9 | Chair transfer |
| 10 | Toilet transfer |
| 11 | Tub transfer |
| 12 | Walk |
| 13 | Stairs |
| Domain 3: cognition | |
| (maximum = 35) | |
| 14 | Comprehension |
| 15 | Expression |
| 16 | Social interaction |
| 17 | Problem solving |
| 18 | Memory |
| Total scores $= 126$ | |

| 7 = Fully independent<br>6 = Modified independent | Unaided |
|---|---|
| 5 = Surveillance is required<br>4 = Minimal aid (75% of children)<br>3 = Moderate help (50% of children) | Helped / Modified Dependent |
| 2 = Maximum help (25% of children)<br>1 = Full help ( <less 25%="" children="" do)<="" of="" td="" than=""><td>Totally Dependent</td></less> | Totally Dependent |

# **Gross Motor Function Measure-88 (Please mark)**

| 1 | A: LYING & ROLLING | | S | CORE | | | |
|---|---|---|---|---|---|---|---|
| 1. | SUP, HEAD IN MIDLINE: TURNS HEAD WITH EXTREMITIES SYMMETRICAL | 0 | 1 | | 2 | 3□ | |
| 2. | SUP: BRINGS HANDS TO MIDLINE, FINGERS ONE WITH THE OTHER | 0 | ] 1 | | 2□ | 3□ | |
| 3. | SUP: LIFTS HEAD 45° | 0 | ] 1 | | 2 | 3□ | |
| 4. | SUP: FLEXES R HIP & KNEE THROUGH FULL RANGE | 0 | 1 | | $_2\square$ | 3□ | |
| 5. | SUP: FLEXES L HIP & KNEE THROUGH FULL RANGE | 0 | ] 1 | | 2 | 3□ | |
| 6. | SUP: REACHES OUT WITH R ARM, HAND CROSSES MIDLINE TOWARD TOY | 0 | ] 1 | | 2 | 3□ | |
| 7. | SUP: REACHES OUT WITH L ARM, HAND CROSSES MIDLINE TOWARD TOY | 0 | ] 1 | | 2 | 3□ | |
| 8. | SUP: ROLLS TO PR OVER R SIDE | 0 | ] 1 | | 2□ | 3□ | |
| 9. | SUP: ROLLS TO PR OVER L SIDE | 0 | ] 1 | | 2 | 3□ | |
| 10. | PR: LIFTS HEAD UPRIGHT | 0 | 1 | | $_2\square$ | 3□ | |
| 11. | PR ON FOREARMS: LIFTS HEAD UPRIGHT, ELBOWS EXT., CHEST RAISED | 0 | ] 1 | | $_2\square$ | $_3\square$ | |
| 12. | problem:probl | oΓ | ] 1 | | $_{2}\square$ | 3□ | |
| 13. | PR ON FOREARMS: WEIGHT ON L FOREARM, FULLY EXTENDS OPPOSITE ARM FORWARD | 0 | ] 1 | | 2 | 3□ | |
| 14. | PR: ROLLS TO SUP OVER R SIDE | 0 | 1 | | $_{2}\square$ | 3□ | |
| 15. | PR: ROLLS TO SUP OVER L SIDE | 0 | ] 1 | | $_{2}\square$ | 3□ | |
| 16. | PR: PIVOTS TO R 90° USING EXTREMITIES | 0 | ] 1 | | 2 | 3□ | |
| 17. | PR: PIVOTS TO L 90° USING EXTREMITIES | ٥ | ] 1 | | $_{2}\square$ | $_3\square$ | |
| | TOTAL DIMENSION A | Г | | | | | 1 |
| | B: SITTING | _ | 8 | CORE | | | _ |
| 18. | SUP, HANDS GRASPED BY EXAMINER: PULLS SELF TO SITTING WITH HEAD CONTROL | ٥ | | | 2 | 3 | |
| 19. | SUP: ROLLS TO R SIDE, ATTAINS SITTING | 0 | | _ | 2<br>2 | 3□ | |
| 20. | SUP: ROLLS TO L SIDE. ATTAINS SITTING | 0 | | | 2<br>2 | 3 | |
| 20. | SIT ON MAT, SUPPORTED AT THORAX BY THERAPIST: LIFTS HEAD UPRIGHT, | 0_ | - 1 | _ | 2 | 30 | |
| 21. | MAINTAINS 3 SECONDS | 0 | 1 | | 2 | 3□ | |
| | SIT ON MAT. SUPPORTED AT THORAX BY THERAPIST: LIFTS HEAD MIDLINE. MAINTAINS | | | _ | _ | _ | |
| 22. | 10 SECONDS | 0 | 1 | | 2 | 3 | |
| 00 | OT OUT A DAY OF PROPERTY OF | | | _ | | | |
| 23. | SIT ON MAT, ARM(S) PROPPING: maintains, 5 seconds | | 0 | 1 | | | 3 |
| 24. | SIT ON MAT: MAINTAIN, ARMS FREE, 3 SECONDS | •••• | $_{0}\square$ | 1 | ] 2 | | 3□ |
| 25. | SIT ON MAT WITH SMALL TOY IN FRONT: LEANS FORWARD, TOUCHESTOY, RE-ERECTS WITHOUT ARM PROPPING | | 0 | 1□ | ] 2 | | 3□ |
| 26 | | | | | 1 | | |
| 26. | SIT ON MAT: TOUCHES TOY PLACED 45° BEHIND CHILD'S R SIDE, RETURNS TO START | | _ | | | | 3 |
| 27. | SIT ON MAT: TOUCHES TOY PLACED 45° BEHIND CHILD'S L SIDE, RETURNS TO START | | 0 | 1 | | | 3 |
| 28. | R SIDE SIT: MAINTAINS, ARMS FREE, 5 SECONDS | | $_{0}\square$ | 1 | ] 2 | | 3□ |
| 29. | L SIDE SIT: MAINTAINS, ARMS FREE, 5 SECONDS | | $_{0}\square$ | 1 | ] 2 | | 3□ |
| 30. | SIT ON MAT: LOWERS TO PR WITH CONTROL | | $_{0}\square$ | 1 | ] 2 | | 3□ |
| 31. | SIT ON MAT WITH FEET IN FRONT: ATTAINS 4 POINT OVER R SIDE | | $\Box_0$ | 1□ | ] 2 | | 3□ |
| 32. | SIT ON MAT WITH FEET IN FRONT: ATTAINS 4 POINT OVER L SIDE | | 0 | 1 | ] 2 | | 3 |
| 33. | SIT ON MAT: PIVOTS 90°, WITHOUT ARMS ASSISTING | | 0 | 1 | | | 3 |
| 34. | SIT ON BENCH: MAINTAINS, ARMS AND FEET FREE, 10 SECONDS | | 0 | 1 | | | 3 |
| 35. | STD: ATTAINS SIT ON SMALL BENCH | | _ | - | _ | | |
| | | | 0 | 1 | | | 3 |
| 36. | ON THE FLOOR: ATTAINS SIT ON SMALL BENCH | | 0 | 1 | | | 3 |
| 37. | ON THE FLOOR: ATTAINS SIT ON LARGE BENCH | | 0 | 1 | 2 | | 3 |
| | TOTAL DIMENSION R | | | | $\neg$ | | |

| Ite | m | C: CRAWLING & KNEELING | | SC | ORE | | NT |
|---|---|---|---|---|---|---|---|
| | 38. | PR: CREEPS FORWARD 1.8m (6') | 0 | 10 | 2 | 3□ | 38. |
| * | 39. | 4 POINT: MAINTAINS, WEIGHT ON HANDS AND KNEES, 10 SECONDS | 0 | 1 | 2 | 3□ | 39. |
| * | 40. | 4 POINT: ATTAINS SIT ARMS FREE | $_{0}\square$ | 1 | 2 | 3□ | 40. |
| * | 41. | PR: ATTAINS 4 POINT, WEIGHT ON HANDS AND KNEES | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 41. |
| * | 42. | 4 POINT: REACHES FORWARD WITH R ARM, HAND ABOVE SHOULDER LEVEL | $_{0}\square$ | 1 | 2 | 3□ | 42. |
| * | 43. | 4 POINT: REACHES FORWARD WITH L ARM, HAND ABOVE SHOULDER LEVEL | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 43. |
| * | 44. | 4 POINT: CRAWLS OR HITCHES FORWARD 1.8m(6') | $_{0}\square$ | 1 | 2 | 3□ | 44. |
| * | 45. | 4 POINT: CRAWLS RECIPROCALLY FORWARD 1.8m ( 6') | $\Box_0$ | 1 | 2 | 3□ | 45. |
| * | 46. | 4 POINT: CRAWLS UP 4 STEPS ON HANDS AND KNEES/FEET | $_{0}\square$ | 1 | 2 | 3□ | 46. |
| | 47. | 4 POINT: CRAWLS BACKWARDS DOWN 4 STEPS ON HANDS AND KNEES/FEET | 0 | 1 | 2 | 3□ | 47. |
| * | 48. | SIT ON MAT: ATTAINS HIGH KN USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | 0 | 1 | 2 | 3□ | 48. |
| | 49. | HIGH KN: ATTAINS HALF KN ON R KNEE USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | 0 | 1 | 2 | 3□ | 49. |
| | 50. | HIGH KN: ATTAINS HALF KN ON L KNEE USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 50. |
| * | 51. | HIGH KN: KN WALKS FORWARD 10 STEPS, ARMS FREE | $\Box_0$ | 1 | 2 | 3□ | 51. |
| TOTAL DIMENSION C | | | | | | | |

| Item | D: STANDING | | SCC | DRE | | NT |
|---|---|---|---|---|---|---|
| * 52 | ON THE FLOOR: PULLS TO STD AT LARGE BENCH | 0 | 1 | 2 | 3□ | 52. |
| * 53 | STD: MAINTAINS, ARMS FREE, 3 SECONDS | 0 | 1 | 2 | 3□ | 53. |
| * 54 | STD: HOLDING ON TO LARGE BENCH WITH ONE HAND, LIFTS R FOOT, 3 SECONDS | 0 | 1 | 2 | 3□ | 54. |
| * 55 | STD: HOLDING ON TO LARGE BENCH WITH ONE HAND, LIFTS L FOOT, 3 SECONDS | 0 | 1 | 2 | 3□ | 55. |
| * 56 | STD: MAINTAINS, ARMS FREE, 20 SECONDS | 0 | 1 | 2 | 3□ | 56. |
| * 57 | STD: LIFTS L FOOT, ARMS FREE, 10 SECONDS | 0 | 1 | 2 | 3□ | 57. |
| * 58 | STD: LIFTS R FOOT, ARMS FREE, 10 SECONDS | 0 | 1 | 2 | 3□ | 58. |
| * 59 | SIT ON SMALL BENCH: ATTAINS STD WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 59. |
| * 60 | HIGH KN: ATTAINS STD THROUGH HALF KN ON R KNEE, WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 60. |
| * 61 | HIGH KN: ATTAINS STD THROUGH HALF KN ON L KNEE, WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 61. |
| * 62 | STD: LOWERS TO SIT ON FLOOR WITH CONTROL, ARMS FREE | 0 | 1 | 2 | 3□ | 62. |
| * 63 | STD: ATTAINS SQUAT, ARMS FREE | 0 | 1 | 2 | 3□ | 63. |
| * 64 | STD: PICKS UP OBJECT FROM FLOOR, ARMS FREE, RETURNS TO STAND | 0 | 1 | 2 | 3 | 64. |
| | TOTAL DIMENSION D | | | | | |

| Item | | E: WALKING, RUNNING & JUMPING | | SCOR | E | | NT |
|---|---|---|---|---|---|---|---|
| * | 65. | STD, 2 HANDS ON LARGE BENCH: CRUISES 5 STEPS TO R | 0 | 1 | 2 | 3□ | 65. |
| * | 66. | STD, 2 HANDS ON LARGE BENCH: CRUISES 5 STEPS TO L | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 66. |
| * | 67. | STD, 2 HANDS HELD: WALKS FORWARD 10 STEPS | $_{0}\square$ | 1 | 2 | 3□ | 67. |
| * | 68. | STD, 1 HAND HELD: WALKS FORWARD 10 STEPS | $_{0}\square$ | 1 | 2 | 3□ | 68. |
| * | 69. | STD: WALKS FORWARD 10 STEPS | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 69. |
| * | 70. | STD: WALKS FORWARD 10 STEPS, STOPS, TURNS 180°, RETURNS | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 70. |
| * | 71. | STD: WALKS BACKWARD 10 STEPS | 0 | 1 | 2 | 3□ | 71. |
| * | 72. | STD: WALKS FORWARD 10 STEPS, CARRYING A LARGE OBJECT WITH 2 HANDS | $_{0}\square$ | 1 | 2 | 3 | 72. |
| * | 73. | STD: WALKS FORWARD 10 CONSECUTIVE STEPS BETWEEN PARALLEL LINES 20cm (8")APART | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 73. |
| * | 74. | STD: WALKS FORWARD 10 CONSECUTIVE STEPS ON A STRAIGHT LINE 2cm (3/4") WIDE | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 74. |
| * | 75. | STD: STEPS OVER STICK AT KNEE LEVEL, R FOOT LEADING | $_{0}\square$ | 1 | 2 | 3□ | 75. |
| * | 76. | STD: STEPS OVER STICK AT KNEE LEVEL, L FOOT LEADING | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 76. |
| * | 77. | STD: RUNS 4.5m (15'), STOPS & RETURNS | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 77. |
| * | 78. | STD: KICKS BALL WITH R FOOT | $_{0}\square$ | 1 | 2 | 3□ | 78. |
| * | 79. | STD: KICKS BALL WITH L FOOT | $_{0}\square$ | 1 | 2 | 3□ | 79. |
| * | 80. | STD: JUMPS 30cm (12") HIGH, BOTH FEET SIMULTANEOUSLY | $_{0}\square$ | 1 | 2 | 3□ | 80. |
| * | 81. | STD: JUMPS FORWARD 30 cm (12"), BOTH FEET SIMULTANEOUSLY | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 81. |
| * | 82. | STD ON R FOOT: HOPS ON R FOOT 10 TIMES WITHIN A 60cm (24") CIRCLE | $_{0}\square$ | 1 | 2 | 3□ | 82. |
| * | 83. | STD ON L FOOT: HOPS ON L FOOT 10 TIMES WITHIN A 60cm (24") CIRCLE | $_{0}\square$ | 1 | 2 | 3□ | 83. |
| * | 84. | STD, HOLDING 1 RAIL: WALKS UP 4 STEPS, HOLDING 1 RAIL, ALTERNATING FEET | $_{0}\square$ | 1 | $_{2}\square$ | 3□ | 84. |
| * | 85. | STD, HOLDING 1 RAIL: WALKS DOWN 4 STEPS, HOLDING 1 RAIL, ALTERNATING FEET | $_{0}\square$ | 1 | 2 | 3□ | 85. |
| * | 86. | STD: WALKS UP 4 STEPS, ALTERNATING FEET | $_{0}\square$ | 1 | 2 | 3□ | 86. |
| * | 87. | STD: WALKS DOWN 4 STEPS, ALTERNATING FEET | $_{0}\square$ | 1 | 2 | 3□ | 87. |
| * | 88. | STD ON 15cm (6") STEP: JUMPS OFF, BOTH FEET SIMULTANEOUSLY | 0 | 1 | 2 | 3□ | 88. |

| TOTAL DIMENSION E |
|-------------------|
|-------------------|